CLINICAL TRIAL: NCT05319301
Title: Identification and Clinical Relevance of an Oxytocin Deficient State Following Melatonin Administration in Patients With Hypopituitarism: a Proof-of-concept, Physiopathological Study With a Control Group
Brief Title: Identification and Clinical Relevance of an Oxytocin Deficient State (Melatonin Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IIBSP-OXI-2021-112
Record Dates: First submitted 2022-03-17; First posted 2022-04-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-03

CONDITIONS: Oxytocin Deficiency; Hypopituitarism; Hypothalamic Obesity; Pituitary Dysfunction; Central Diabetes Insipidus; Social Isolation
Keywords: oxytocin; melatonin; hypopituitarism; vasopresin deficiency
MeSH Terms: conditions — Hypopituitarism; Sexual Infantilism; Diabetes Insipidus, Neurogenic; Social Isolation | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with hypopituitarism (Experimental): A single dose of melatonin administration
  Interventions: Dietary Supplement: Melatonin
- Healthy controls (Active Comparator): A single dose of melatonin administration
  Interventions: Dietary Supplement: Melatonin

INTERVENTIONS:
Dietary Supplement: Melatonin — A single dose of melatonin (1.9 mg)

SUMMARY:
Oxytocin (OT) is a hypothalamic peptide that enters the peripheral circulation via the posterior pituitary gland. OT plays a key role in regulating appetite, psychopathology, prosocial behavior and sexual function. Hypopituitarism is associated with increased obesity, increased psychopathology, sexual and prosocial dysfunction despite appropriate hormone replacement. A few studies suggest the existence of a possible OT deficient state in hypopituitarism. In animal models, melatonin has shown to increase OT release.

This study is designed to evaluate oxytocin values after administration of melatonin in adults (healthy volunteers and patients with hypopituitarism).

The investigators hypothesize that OT response will be blunted following melatonin in patients with hypopituitarism compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypopituitarism (HYPO) (>1 pituitary hormone deficiency) and stable hormone replacement for the prior three months
* At least one clinical sign of hypothalamic damage

Exclusion Criteria:

* uncorrected hormone deficiency
* creatinine >1.5mg/dL
* alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5x upper limit of normal
* hematocrit less than 30%
* suicidality or active psychosis
* participation in a trial with investigational drugs within 30 days
* using a high glucocorticoid dose
* vigorous physical exercise
* alcohol intake within 24 hours before the study participation
* evidence of any acute illness or any illness that the Investigator determines could interfere with study participation or safety
* pregnancy or breastfeeding for last 8 weeks
* known allergies towards melatonin
* patients refusing or unable to give written informed consent
* patients receiving fluvoxamine and/or impossibility to stop hypnotics 48 hours prior to the study visit.
* Additionally for healthy controls: the presence of brain or pituitary tumor, radiation involving the hypothalamus or pituitary, history of hypopituitarism or receiving testosterone or glucocorticoids esters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change in oxytocin concentration | Baseline blood exam (timepoint 0) and further blood collections after 30, 60, 90 and 120 minutes after baseline blood collection
  Change in oxytocin concentration (pg/mL) after administration of 1.9 mg of melatonin orally.

SECONDARY OUTCOMES:
Maximal change in oxytocin concentration (pg/mL) | Within the two hours after the injection
  Maximal change in oxytocin concentration (pg/mL) after administration of 1.9 mg of melatonin administered orally.
Overall oxytocin secretion | Within the two hours after the injection
  Oxytocin area under the curve after administration of 1.9 melatonin administered orally
Mood assessment | At baseline
  Correlation between Beck Depression Inventory-2 score (range from 0 to 63, higher scores mean a worse outcome) and baseline oxytocin concentration (pg/mL)
Quality of life assessment | At baseline
  Correlation between 36 item- Short Form Health Survey score (range from 0 to 100, the higher scores indicate better health status) and baseline oxytocin concentration (pg/mL)
Impulsivity assessment | At baseline
  Correlation between Barratt Impulsiveness Scale (range from 30 to 120, higher scores indicate greater impulsivity) and baseline oxytocin concentration (pg/mL)
Alexithymia assessment | At baseline
  Correlation between Toronto Alexithymia scales-20 score (range from 20 to 100, higher scores mean a worse outcome) and baseline oxytocin concentration (pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain